CLINICAL TRIAL: NCT03018821
Title: Efficacy Comparison Between Two Kind of Chinese Herbal Formulas on Traditional Chinese Medicine Syndromes Among Chronic Hepatitis Patients
Brief Title: The Study of Two Different Chinese Traditional Medicine Treatment on Chronic Hepatitis B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Traditional Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XAZYYLS2017-02
Record Dates: First submitted 2017-01-06; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis B， Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir

ARMS (3):
- Standard CMF (Active Comparator): Standard Chinese medical formulas (CMF) for the corresponding TCM syndromes, plus an anti-virus treatment of western drugs (such as Entecavir or Tenofovir).
  1. Yinchengao Decoction plus Ganlu Detoxification Pill for the Traditional Chinese Medicine (TCM) syndrome: Damp-heat blocking middle jiao
  2. Chaihu Shugan San for the TCM syndrome: Liver depression and qi stagnation
  3. Xiaoyao powder for the TCM syndrome: Stagnation of liver qi and spleen deficiency.
  4. Yiguan Decoction for the TCM syndrome: Yin deficiency of liver and kidney
  5. Fuzilizhong Decoction plus Jinkui Shenqi Bolus for the TCM syndrome: Yang deficiency of spleen and kidney
  6. Ge Xia Zhu Yu Decoction for the TCM syndrome: Internal blood stasis
  Interventions: Drug: Standard - Yinchengao Decoction plus Ganlu Detoxification Pill; Drug: Entecavir or Tenofovir; Drug: Standard - Ge Xia Zhu Yu Decoction; Drug: Standard - Chaihu Shugan San; Drug: Standard - Xiaoyao powder; Drug: Standard - Yiguan Decoction; Drug: Standard - Fuzilizhong Decoction plus Jinkui Shenqi Bolus
- Advanced CMF (Experimental): Advanced TCM formulas for corresponding TCM syndromes provided by famous TCM doctors who were national wide known in China, plus an anti-virus western drugs (such as Entecavir or Tenofovir).
  1. Taohong Huazhuo Decoction for the Traditional Chinese Medicine (TCM) syndrome: Damp-heat blocking middle jiao
  2. Soothe the liver and regulate qi Decoction for the TCM syndrome: Liver depression and qi stagnation
  3. Supplemented Ganbi Decoction for the TCM syndrome: Stagnation of liver qi and spleen deficiency.
  4. Supplemented Zimu Dan for the TCM syndrome: Yin deficiency of liver and kidney
  5. Guifu Erxian Decoction for the TCM syndrome: Yang deficiency of spleen and kidney
  6. Supplemented Ganji Decoction for the TCM syndrome: Internal blood stasis
  Interventions: Drug: Entecavir or Tenofovir; Drug: Advanced - Supplemented Taohong Huazhuo Decoction; Drug: Advanced - Soothe the liver and regulate qi Decoction; Drug: Advanced - Supplemented Ganbi Decoction; Drug: Advanced - Supplemented Zimu Dan; Drug: Advanced - Guifu Erxian Decoction; Drug: Advanced - Supplemented Ganji Decoction
- Pure Entecavir or Tenofovir (Experimental): Use an anti-virus western drug alone (such as Entecavir or Tenofovir).
  Interventions: Drug: Entecavir or Tenofovir

INTERVENTIONS:
Drug: Standard - Yinchengao Decoction plus Ganlu Detoxification Pill — Yinchengao Decoction plus Ganlu Detoxification Pill is one Chinese Medicine Formula for the TCM syndrome: Damp-heat blocking middle jiao.
  Arms: Standard CMF
Drug: Entecavir or Tenofovir — Western drug for anti-HBV such as Entecavir and Tenofovir
Drug: Standard - Ge Xia Zhu Yu Decoction — Ge Xia Zhu Yu Decoction is one Chinese Medicine Formula for the TCM syndrome: internal blood stasis.
  Arms: Standard CMF
Drug: Advanced - Supplemented Taohong Huazhuo Decoction — Supplemented Taohong Huazhuo Decoction is one Chinese Medicine Formula suggested by national wide known TCM doctors who expertise in chronic hepatitis B for the TCM syndrome: Damp-heat blocking middle jiao.
  Arms: Advanced CMF
Drug: Standard - Chaihu Shugan San — Chaihu Shugan San is one Chinese Medicine Formula for the TCM syndrome: Liver depression and qi stagnation.
  Arms: Standard CMF
Drug: Advanced - Soothe the liver and regulate qi Decoction — Soothe the liver and regulate qi Decoction is one Chinese Medicine Formula suggested by national wide known TCM doctors who expertise in chronic hepatitis B for the TCM syndrome: Liver depression and qi stagnation.
  Arms: Advanced CMF
Drug: Standard - Xiaoyao powder — Xiaoyao powder is one Chinese Medicine Formula for the TCM syndrome: Stagnation of liver qi and spleen deficiency.
  Arms: Standard CMF
Drug: Advanced - Supplemented Ganbi Decoction — Supplemented Ganbi Decoction is one Chinese Medicine Formula suggested by national wide known TCM doctors who expertise in chronic hepatitis B for the TCM syndrome: Stagnation of liver qi and spleen deficiency.
  Arms: Advanced CMF
Drug: Standard - Yiguan Decoction — Yiguan Decoction is one Chinese Medicine Formula for the TCM syndrome: Yin deficiency of liver and kidney.
  Arms: Standard CMF
Drug: Advanced - Supplemented Zimu Dan — Supplemented Zimu Dan is one Chinese Medicine Formula suggested by national wide known TCM doctors who expertise in chronic hepatitis B for the TCM syndrome: Yin deficiency of liver and kidney.
  Arms: Advanced CMF
Drug: Standard - Fuzilizhong Decoction plus Jinkui Shenqi Bolus — Fuzilizhong Decoction plus Jinkui Shenqi Bolus is one Chinese Medicine Formula for the TCM syndrome: Yang deficiency of spleen and kidney.
  Arms: Standard CMF
Drug: Advanced - Guifu Erxian Decoction — Guifu Erxian Decoction is one Chinese Medicine Formula suggested by national wide known TCM doctors who expertise in chronic hepatitis B for the TCM syndrome: Yang deficiency of spleen and kidney.
  Arms: Advanced CMF
Drug: Advanced - Supplemented Ganji Decoction — Supplemented Ganji Decoction is one Chinese Medicine Formula suggested by national wide known TCM doctors who expertise in chronic hepatitis B for the TCM syndrome: internal blood stasis.
  Arms: Advanced CMF

SUMMARY:
Although the incidence of Hepatitis B has been decreased a lot recently years, there are still quite a few chronic hepatitis B patients in China. The anti-virus drugs of western medicine such as Entecavir and Tenofovir have been proved effective on decreasing the serum hepatitis B virus (HBV) level, on the other hand, Chinese materia medica showed effective on TCM syndromes of chronic hepatitis B (CHB) such as hypochondriac pain, jaundice and abdominal mass. Besides, the hepatic fibrosis could be delayed after the appropriate treatment of TCM. This study is a multicenter, randomized, open label, parallel group clinical trial to evaluate the efficacy of two different traditional Chinese medicine (TCM) herbal treatment on chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* 18<=age at treatment<=65 years old
* Was diagnosed as chronic hepatitis B (ICD10:K73.901) and one of the following Chinese syndromes: hypochondriac pain (TCD:BNG010), jaundice(TCD:BNG020) or abdominal mass (TCD:BNG040).

Exclusion Criteria:

* Combined with other virus hepatitis or alcoholic hepatitis
* Combined with autoimmune disease
* Combined with liver cancer or cirrhosis
* Combined with severe hepatitis with or without complications
* Combined with unstable cardio-cerebrovascular disease
* Combined with severe lung, kidney, endocrine system, nervous system and hematological system diseases
* Combined with Tuberculosis
* Chronic hepatitis patients with ongoing INF treatment
* Woman with pregnancy or breasting feeding
* Mental disorder and can not express self clearly
* Cannot speak Chinese
* Allergic constitution or allergy to multiple drugs
* Refuse to enroll into the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Traditional Chinese Medicine symptom scale | Change of TCM symptom scale between baseline and sixth months of treatment

SECONDARY OUTCOMES:
The change of liver fibrosis | Chnage of liver fibrosis between baseline and 6th months of treatment
  Use change of FibroScan measurement of liver between baseline and 6th months of treatment to express the change of liver fibrosis
Overall effectiveness of treatment defined by the guidelines for prevention and treatment of chronic hepatitis B | Overall effectiveness of treatment between baseline and 6th months of treatment
  Treatments were completely effective, partially effective or not effective after treatment.
  Complete effective: Alanine aminotransferase normal, HBV DNA, HBeAg and HBsAg are negative
  Partially effective: Alanine aminotransferase normal, HBV DNA, HBeAg are negative and HBsAg stay positive
  Not effective: Did not reach any one of what are listed above.

CONTACTS AND LOCATIONS:
Locations (1):
- Xi'an Traditional Medicine Hospital, Xi'an, Shaanxi, China